CLINICAL TRIAL: NCT02075346
Title: Sensor Off Studies Using a Nellcor Bedside Respiratory Patient Monitoring System, Configured With the Multi-functional Respiratory PCBA
Brief Title: Bedside Respiratory Patient Monitoring System - Sensor Off Study
Acronym: BRPMS
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: COVMOPR0419
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2013-12

CONDITIONS: Healthy Volunteers
Keywords: Patient safety monitors

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

SUMMARY:
Use of an investigational oximetry system to evaluate the triggering of the "sensor off" status with the marketed off-the-shelf sensors.

DETAILED DESCRIPTION:
The Multi-functional Patient Monitoring PCBA is an electronic circuit board in the monitoring system that performs calculations.

The study will evaluate the performance of the Sensor Off New Patient Monitoring system by exposing the sensor to an ambient light source, sensor slipping off the finger with the light emitter and detector facing each other or a sensor slipping off under a blanket.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18 years or older (inclusive)
* Subject is able to participate for the duration of the study
* Subject is willing to sign an informed consent

Exclusion Criteria:

* Previous injury or trauma to fingers or hands that may change blood flow or vascular supply and affect our ability to test sensors.
* Physiologic abnormalities that prevent proper application of pulse oximetry sensor.
* Severe contact allergies that cause a reaction to standard adhesive materials such as those found in medical sensors and electrodes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 20 subjects recruited from the Clinical Laboratory subject data base.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2013-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
To validate that the device posts a "Sensor Off" message within one minute after the sensor is removed at least ninety percent of the time. | The planned duration of the study is 1 month.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Kelley, MD, Principal Investigator — Medtronic - MITG
Locations (1):
- Boulder Clinical Laboratory, Boulder, Colorado, United States